CLINICAL TRIAL: NCT03789929
Title: Scientific Evaluation of Online-Trainings for Emotional Competence, Compassion and Relationship Competences
Brief Title: Emotional Competence and Compassion Online-Training
Acronym: ECCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Principal Investigator, Charite University, Berlin, Germany
Other Study IDs: ECCO
Record Dates: First submitted 2018-12-14; First posted 2018-12-31 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Emotional Intelligence
Keywords: Stress; Emotion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The Emotional Backpack: Healthy adults participating in the offered online-course on their own initiative.
  Interventions: Behavioral: The Emotional Backpack
- Feelings as Powers: Healthy adults participating in the offered online-course on their own initiative.
  Interventions: Behavioral: Feelings as Powers

INTERVENTIONS:
Behavioral: The Emotional Backpack — In this 4 weeks course participants learn how to process difficult emotions that has been overwhelming in the past. They learn how they can use the support of other people and support other people in the processing emotions within a simple and easy to learn setting.
  Groups: The Emotional Backpack
Behavioral: Feelings as Powers — In this 3 months course participants learn about the empowering potential of their feelings as well as the difficult aspects of them. In addition to that they learn techniques how to deal with difficult emotions.
  Groups: Feelings as Powers

SUMMARY:
In this study two different online-courses about emotional competence and compassion are scientifically evaluated with psychometric questionnaires and heart rate variability measuring.

DETAILED DESCRIPTION:
Stress and stress related diseases are becoming a huge health burden in modern societies. Psycho-emotional stress plays a key role in stress regulation. Therefore this study aims to investigate the effects of online-courses addressing emotion regulation.

For this aim several different online-courses about emotional competence and compassion are scientifically evaluated with psychometric questionnaires and heart rate variability measuring. The courses are planned by the trainers and people register on their own initiative.

The courses have a duration of 4 weeks or three months. They consist of video lectures that explain the content as well as videos giving exercises about the character of the different feelings and about the characteristics of emotions. They teach practices on how to use feelings as an empowering force in life and how to deal with difficult emotions.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years
* participation in one of the included courses
* e-mail address

Exclusion Criteria:

* participation in another study
* no verbal communication (german) possible
* dementia or another disease that limits cognitive abilities

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy adults who enrolled themselves from their own initiative into one of the included courses
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Self-Report Measure for the Assessment of Emotion Regulation Skills (SEK-27) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 0-108, higher score meaning a better outcome

SECONDARY OUTCOMES:
Saarbrücken Personality Questionnaire (SPF) based on the Interpersonal Reactivity Index (IRI) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 16-80, higher score meaning a better outcome
The World Health Organisation- Five Well-Being Index (WHO-5) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 0-100, higher score meaning a better outcome
General Self-efficacy Short Scale (ASKU) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 3-15, higher score meaning a better outcome
Hospital Anxiety and Depression Scale (HADS) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 0-42, lower score meaning a better outcome
Mindful Attention Awareness Scale (MAAS) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 15-90, higher score meaning a better outcome
Perceived Stress Scale (PSS-10) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 0-40, lower score meaning a better outcome
Medical Outcomes Study Short Form (MOS SF-36) | Assessing change from baseline to 3 months and 6 months after baseline in single workshops and baseline to 3, 6, 9 and 12 months after baseline in the yearly program
  Assessing full scale, range 0-100, higher score meaning a better outcome
Heart Rate Variability (HRV) | Assessing change from baseline to 3 and 6 months after baseline in the yearly program
  24h measuring

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, prof. Dr., Principal Investigator — Charite - Universitätsmedizin Berlin
Locations (1):
- Charité Medical University, Department of Integrative Medicine at the Immanual Hospital Berlin, Berlin-Zehlendorf, State of Berlin, Germany